CLINICAL TRIAL: NCT07133074
Title: Optimizing Antibiotic Selection in Hematologic Malignancy Patients With Reported Beta-lactam Allergy - Intervention
Brief Title: Allergy Delabeling in Antibiotic Stewardship - Intervention
Acronym: RENEW-IN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ebbing Lautenbach (Other)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor-Investigator, Ebbing Lautenbach, Professor of Medicine and Epidemiology, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 855861; R01HS029879 (AHRQ)
Record Dates: First submitted 2025-06-16; First posted 2025-08-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Beta Lactam Allergy; Hematologic Malignancy
Keywords: penicillin allergy; hematologic cancer; allergy delabeling
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Interrupted Time Series Analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients who enroll in the RENEW intervention (Other): Patients who agree to actively participate in the RENEW intervention designed to identify opportunities to have the beta lactam allergy label removed from their electronic medical record.
  Interventions: Diagnostic Test: RENEW-IN Algorithm for assessment of a beta-lactam intervention
- Patients hospitalized with a hematologic malignancy in the time period prior to the intervention (Other): Patients who are hospitalized with a hematologic malignancy who would meet the inclusion criteria for the intervention but who were not approached since they were hospitalized in the time period prior to introduction of the intervention. These patients will be used as a control group. Charts for these patients will be retrospectively reviewed and data will be extracted for analysis of the primary and secondary outcomes.
  Interventions: Other: EMR Review

INTERVENTIONS:
Diagnostic Test: RENEW-IN Algorithm for assessment of a beta-lactam intervention — The RENEW-IN intervention includes a detailed assessment of the participant's beta-lactam allergy history and determination of a risk-level for allergy-delabeling.
  Arms: Patients who enroll in the RENEW intervention
Other: EMR Review — Electronic medical record review for comparative analysis
  Arms: Patients hospitalized with a hematologic malignancy in the time period prior to the intervention

SUMMARY:
The overall goal of the RENEW-IN intervention is to assess the impact of a BL allergy delabeling intervention on antibiotic use and clinical outcomes in patients with a hematologic malignancy.

DETAILED DESCRIPTION:
The RENEW clinical intervention is designed to evaluate the impact of a comprehensive beta lactam allergy delabeling intervention on clinical outcomes among patients hospitalized with a hematologic malignancy (HM).

HM patients are at a high risk of infection-related complications but are limited to antibiotic therapy based on self-reported allergies.

Beta-lactam (BL) antibiotics are a preferred treatment option for many bacterial infections, however, these antibiotics remain inaccessible as a treatment option for patients with a self-reported BL allergy. In the hospital setting, BL allergies are documented in the electronic medical record in up to 20% of hospitalized patients. Prior studies have shown that 90% of the patients for whom these allergies are reported are able to tolerate penicillin (PCN) or other BLs. Delabeling strategies to correctly identify true BL allergies in the general hospital population have proven successful. However, these studies have not been conducted among patients diagnosed with a hematological malignancy. The investigators propose to test the impact of a pharmacist-led BL allergy delabeling intervention on clinical outcomes and antibiotic use in hospitalized patients with HM.

The intervention is a multi-step PCN delabeling strategy that includes 1) an assessment of the participant's BL allergy by a clinical pharmacist based on a detailed medical history; 2) assignment of additional allergy testing based on the RENEW-IN algorithm; and 3) delabeling of the allergy within the participants electronic medical record if appropriate.

ELIGIBILITY:
Inclusion Criteria:

* all patients with a hematologic malignancy (including Hodgkin and non-Hodgkin lymphoma, leukemia, and myeloma) admitted to an inpatient oncology service
* reported history of a beta-lactam (BL) allergy (i.e., penicillin, cephalosporin, and/or carbapenem)

Exclusion Criteria:

* patients with a history of severe cutaneous adverse reaction
* patients with a history of Stevens-Johnson syndrome
* patients with a history of toxic epidermal necrolysis
* patients with a history of drug-induced exfoliative dermatitis
* patients with a history of drug reaction with eosinophilia and systemic symptoms
* patients with a history of acute generalized exanthematous pustulosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3800 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Antibiotic Days of therapy | From baseline enrollment to end of index hospitalization or death, up to 36 months
  Proportion of participants prescribed an antibiotic during index hospitalization, from enrollment in the study to hospital discharge or death, whichever occurs first
Hospital length of stay | From baseline enrollment to end of index index hospitalization or death, up to 36 months
  Number of days participants are admitted to the hospital during the index visit, from enrollment in the study to hospital discharge or death, whichever occurs first

SECONDARY OUTCOMES:
Clinical Cultures positive for multi-drug resistant organisms | From baseline enrollment to end of index index hospitalization or death, up to 36 months
  Proportion of participants diagnosed with multi-drug resistant organism during index hospitalization, from enrollment in the study to hospital discharge or death, whichever occurs first
Clinical Cultures positive for Clostridioides difficile infection | From baseline enrollment to end of index index hospitalization or death, up to 36 months
  Proportion of participants diagnosed with Clostridioides difficile infection during index hospitalization, from enrollment in the study to hospital discharge or death, whichever occurs first
Clinical Cultures positive for Health-care Associated Infections (HAIs) | From baseline enrollment to end of index index hospitalization or death, up to 36 months
  Proportion of participants diagnosed during index visit with an infection identified as related to their hospitalization, from enrollment in the study to hospital discharge or death, whichever occurs first
Need for ICU transfer | From baseline enrollment to end of index index hospitalization or death, up to 36 months
  Proportion of participants admitted to the ICU during their index hospitalization, from enrollment in the study to hospital discharge or death, whichever occurs first
ICU length of stay | From baseline enrollment to end of index index hospitalization or death, up to 36 months
  Number of days participants are admitted to the ICU during their index hospitalization, from enrollment in the study to hospital discharge or death, whichever occurs first
Patient Disposition | From baseline enrollment to end of index index hospitalization or death, up to 36 months
  Proportion of participants who are discharged from the hospital at the end of their index visit compared to the number of participants who expire during their index visit